CLINICAL TRIAL: NCT07367139
Title: Occupational Exposure to Whole Body Vibration Among U.S. Military Veterans: Acute and Chronic Contributions to Musculoskeletal Disorders and Spine-Area Pain, and the Role of Water
Brief Title: Occupational Exposure to Whole Body Vibration Among U.S. Military Veterans: Acute and Chronic Contributions to Musculoskeletal Disorders and Spine-Area Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milwaukee VA Medical Center (U.S. Federal Agency)
Collaborators: Medical College of Wisconsin (Other); Indiana University (Other); VA Office of Research and Development (U.S. Federal Agency); Naval Aeromedical Research Unit, Dayton (U.S. Federal Agency)
Responsible Party: Principal Investigator, Brian D. Stemper, Research Health Scientist, Milwaukee VA Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1918913
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Spine Health; Spine Injuries and Disorders; Spine Degeneration; Whole Body Vibration
Keywords: Biomechanics; Magnetic Resonance Imaging (MRI); Whole Body Vibration; Lumbar Spine; Degeneration; Intervertebral Disc; Hydration; Oswestry Disability Index; PainDETECT; Pain Catastrophizing; PROMIS; Brief Pain Inventory; Longitudinal; Endplate
MeSH Terms: conditions — Disease | interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Longitudinal effects of current or prior whole body vibration. (No Intervention): Determine the impact of acute and longitudinal WBV on lumbar spine endplate health. The objective is to perform a repeated measures study using multi-parametric MRI to assess Veteran endplate health. Veterans will participate in pain assessments and MRI scans annually for three years to track the progression of whole body vibration-related changes in the lumbar spine endplates and intervertebral discs. Current and prior whole body vibration characteristics will be correlated to pain scores and MRI changes.
- Determine how lumbar disc fluid flow is acutely affected by whole body vibrati (No Intervention): The objective is to perform a repeated measures study to quantify changes in lumbar spine T2 relaxation times and volumetric MRI data following acute experimental vibrational exposure to determine fluid transport patterns and morphological changes. Veterans will participate in pain questionnaires, and receive Upright MRI scans prior to and immediately following 30 minutes of low magnitude whole body vibration. This unique protocol will allow us to assess acute changes in MR metrics and structural dimensions of the lumbar spine following exposure to WBV by comparing measurements obtained immediately following experimental WBV to pre-WBV measurements.
- Effect of hydration on lumbar spine response to whole body vibration (Experimental): This arm will determine whether individual hydration state influences IVD water dynamics following acute vibrational exposure. The objective is to assess the impact of hydration on IVD fluid distribution and transport in response to acute vibration utilizing multi-parametric MRI analysis. This will allow for evaluation of hydration as a potential factor for rehabilitation, treatment, and prevention of early degeneration related to WBV. MRI scans will be obtained under two conditions: hydrated and dehydrated. For the hydrated MRI scans, research subjects will be asked to consume a minimum of 2.7 liters of fluid per day for three days leading up the MRI date. For the dehydrated MRI scans, research subjects will be asked to consume about 1.3 liters of fluid per day for three days leading up to the MRI date. WBV induced changes to IVD water dynamics will be compared within subjects for the hydration, dehydration and control conditions.
  Interventions: Other: Water

INTERVENTIONS:
Other: Water — Aim 3 will evaluate the effect of hydration and dehydration on acute whole body vibration response of the lumbar spine endplate and intervertebral disc.
  Arms: Effect of hydration on lumbar spine response to whole body vibration

SUMMARY:
Significance to VA: There is a lack of prospective longitudinal studies investigating the relationship between risk factors to Veterans and development and progression of musculoskeletal (MSK) spine injury and pain. Military operational exposure to whole body vibration (WBV) is known to contribute to MSK disorders and pain. Our preliminary studies identified accelerated lumbar and cervical spine degenerative changes in military fighter pilots and helicopter aircrew compared to age- and sex-matched civilian controls. Those changes were likely associated with WBV that military aircrew experience during flight training, primarily affected intervertebral discs (IVDs) and endplates, were associated with neck and back pain symptoms and reduced functional capacity, and are likely to lead to lifelong spine-related issues. Therefore, these aircrew, and other military personnel that experience occupational WBV, are likely to enter the VA Healthcare system with pre-existing degenerative changes and spine-related pain symptoms that can progress over time. Similarly, many Veterans enter civilian occupations that involve WBV such as truck drivers and heavy equipment operators that may also have detrimental effects to the spine and lead to spine-related pain. Development of informed interventions and treatment protocols requires a mechanistic understanding of how the spine is acutely and chronically affected by occupational WBV from both structural and physiological perspectives. Innovation and Impact: Novel multi-parametric application of noninvasive magnetic resonance imaging (MRI) techniques such as arterial spin labeling (ASL), T2* decay from ultra short TE, and diffusion MRI can provide early objective indications of endplate degenerative state and IVD hydration and perfusion, and novel application of upright MR imaging allows for gravitational loading of the IVD while observing segmental and region IVD fluid distribution and transport patterns. Specific Aims: The goal of the proposed effort is to characterize the effects of previous military and current civilian occupational WBV on IVD and endplate health and degeneration (Aim 1), and segmental and regional IVD fluid distribution and transport differences (Aim 2). The endplates contain vasculature that permits IVD fluid exchange and may be linked to IVD fluid dynamics. We propose looking for connections between segmental and regional IVD fluid dynamics, degenerative state of the associated endplates, and WBV exposure (acute-controlled and longitudinal-occupational). Finally, we propose evaluating the impact of body hydration state on IVD fluid distribution and transport following acute (30 min) controlled WBV (Aim 3). Cumulatively, these results inform population-specific preventative measures to preserve endplate health for Veterans in occupations that present with WBV and identify potential areas for further research and targeted treatment of MSK disorders and MSK pain. Methodology: This study will explore acute and chronic changes to the structure and physiology of the spine by enrolling Veterans with prior military or current civilian occupation that involves daily WBV. Advanced MRI sequences will identify endplate sclerosis and physiological changes including disc hydration and perfusion. Acute effects of WBV will be assessed using pre/post MRI scans with experimental WBV. Path to translation/Implementation: Our existing relationships with VA clinicians, including spine surgeons, physical medicine and rehabilitation, and pain medicine, will ensure VA patient applicability of these findings and will help to translate any outcomes from this research and future studies directly into patient care.

DETAILED DESCRIPTION:
Musculoskeletal (MSK) disorders and spine-related pain are major health concerns among veterans. Low back pain is the most common chronic pain condition among Veterans, contributing significantly to healthcare utilization and rising treatment costs within the Veteran's Health Administration (VHA). As VHA community care expenditures more than doubled between 2017 and 2021, the growing demand for chronic pain services underscores the need for improved understanding of the mechanisms that contribute to spine degeneration in this population. There is evidence that occupational exposure to whole body vibration (WBV) is associated with an increased risk for a multitude of negative health outcomes, including MSK pain in the back and neck. However, despite extensive research on low back pain etiology and disc degeneration, major gaps persist around early detection of endplate degeneration and the impact of acute or chronic WBV exposure on IVD health.

The ubiquitous nature of low back pain in the general public but especially in veterans shows that there is a strong medical need for better understanding of the biomechanics of spine health. This study can help clinical practice by identifying early detection biomarkers with non-invasive MRI techniques and to investigate hydration as a protective mechanism.

The problem of low back pain and spine health is especially relevant within veterans because while service members are generally healthier than the typical U.S. adult of similar age at the time they enter service (because of rigorous physical and mental screening requirements to join the military, continued fitness standards, and access to comprehensive healthcare), research has shown that Veterans have poorer overall health-related quality of life than nonveterans and a high prevalence of back pain-related conditions. Veterans have often been exposed to WBV during their military career while in armored or heavy vehicles or in aircraft. Many veterans also continue to be exposed to WBV in their post-military careers with 28.5% working in natural resources, construction and maintenance or production, transportation and material moving. These jobs and many others may expose workers to WBV while operating vehicles (trucks, construction and heavy machinery), or operating tools where the vibrational amplitude is large enough to transmit to the body. These WBV exposures during their military career and post military career carries an increased risk of negative health outcomes including MSK pain in the back and neck.

While we know that many veterans are exposed to these conditions and they are associated with an increased risk of MSK pain, understanding the biomechanics will help understand how to prevent and treat those long term or chronic injuries. These are knowledge gaps that we have identified in relation to intervertebral disc health and exposure to WBV:

1. Segment- and region-specific disc fluid dynamics under WBV are poorly understood.

   While diurnal disc fluid migration patterns have been documented, the impact of acute or chronic WBV on nucleus pulposus and annulus fibrosis fluid distribution, especially across lumbar levels, remains unknown.
2. Early endplate degeneration cannot currently be detected noninvasively. Modic bone marrow changes observable with MRI lack sensitivity and reflect late-stage pathology. No clinical imaging method reliably identifies early degenerative alterations of the cartilaginous or bony endplates.
3. The relationship between endplate health and disc fluid transport under WBV exposure is unclear.

   Endplate degeneration likely disrupts regional fluid exchange and may drive segment-dependent susceptibility to WBV-induced disc injury.
4. No prior studies have integrated advanced quantitative MRI techniques to evaluate endplate perfusion, disc fluid movement, and WBV response.

Although dynamic contrast-enhanced MRI can measure endplate perfusion, concerns about gadolinium retention limit its use. Non-contrast alternatives such as arterial spin labeling (ASL) have not been applied to endplate assessment.

This study will address those gaps by combining multi-parametric MRI and groups selected for both acute and longitudinal occupational exposure to WBV to evaluate IVD fluid transport and endplate health. By addressing these gaps, this study will advance understanding of the biomechanical and physiological impacts of WBV on spine health.

We seek to understand the connection between WBV exposure and spine health by comparing groups of veterans with history of or ongoing exposure to WBV and using advanced MRI techniques to study intervertebral disc (IVD) and vertebral endplate health. We also seek to study the acute changes in IVD and vertebral endplate biology before and after exposure to WBV and whether individual hydration state influences IVD water dynamics.

The specific aims are:

Aim 1: Determine the impact of acute and longitudinal WBV on lumbar spine endplate health.

Aim 2: Determine how segmental lumbar and regional IVD fluid distribution and transport are acutely affected by WBV and determine if there are correlations with endplate health.

Aim 3: Determine whether individual hydration state influences IVD water dynamics following acute vibrational exposure.

We hypothesize the following

Specific Aim 1 Hypothesis 1: Multi-parametric MRI will reveal Veterans with previous military WBV exposure have more degenerative endplate markers when compared to Veterans with no occupational WBV exposure.

Hypothesis 2: Multi-parametric MRI in Veterans with current occupational exposure to WBV, but with no previous military WBV exposure, will have earlier expression of degenerative endplate markers when compared to Veterans with no WBV exposure.

Hypothesis 3: The rate of change for degenerative endplate markers over the four-year duration of the study will be greater for Veterans with current occupational WBV exposure than for Veterans that had previous military occupational WBV exposure.

Specific Aim 2 Hypothesis 1: Veterans who routinely experience occupational WBV will exhibit less IVD regional fluid distribution before and after experimental WBV, while those without daily WBV will have greater changes in IVD regional fluid distribution following experimental WBV, with water moving from the NP into the AF or out of the disc.

Hypothesis 2: Veterans who routinely experience occupational WBV will exhibit a cranial to caudal decrease in water transport as well as a decrease in baseline water distribution.

Hypothesis 3: Degenerative endplate health will be correlated with decreased lumbar spine water distribution and transport.

Specific Aim 3 Hypothesis 1: Participants in a low-hydration state will exhibit a larger reduction in intervertebral disc (IVD) water content and altered fluid-transport metrics after 30 minutes of controlled seated vibration than participants in a normal/high-hydration state.

This research is relevant to the VA due to approximately 50% of veterans experiencing chronic pain with lower back pain being the most common type of chronic pain. This is one of the most common reasons for seeking care within the VHA and this creates a significant financial burden on the Veterans Health Administration. There is also data that shows despite service members being generally healthier than the typical U.S. adult when entering service, there is a high incidence of lower back pain among service members and that veterans have poorer overall health related quality of life than non-veterans. Occupational exposure to vibration is associated with an increased risk for a multitude of negative health outcomes, including MSK pain in the back and neck.

Study Design:

This study will investigate acute and chronic effects of occupational whole-body vibration on the health of lumbar spine endplates and intervertebral discs by studying Veterans that had occupational exposure to WBV in their military occupation and Veterans with current civilian occupations that involve WBV. The approximate study timeline, as outlined in the grant proposal, is shown below. Lumbar spine endplate characteristics and intervertebral disc perfusion and hydration in both study groups will be compared to age- and sex-matched Veteran controls with no history of occupational WBV. The volunteer population will be chosen to represent the ethnic and sex distribution of the Zablocki Veterans Affairs Medical Center patient population. Current and military occupations will be selected to maximize consistency in WBV characteristics. For example, the ZVAMC patient population includes both truck drivers and heavy equipment operators. However, given that the WBV characteristics (e.g., frequency and magnitude of vibration) between those occupations are different, which will likely have different acute and chronic effects on the spine, preference in the research population be given to maximize consistency in the WBV environment across the research subject population. We will follow a similar procedure for choosing Veterans with military occupational WBV. Occupations unique to the military, such as helicopter aircrew, will be given priority although other occupations such as truck drivers, etc. will be targeted if we are not able to enroll Veterans with previous military helicopter occupation in sufficient numbers. The initial questionnaire will also include the Oswestry Disability Index (ODI), which will provide information on the impact of low back pain for each prospective subject's daily activities and function. The ODI will also be used in the selection of subjects for the MRI arm of the study to ensure a consistent sample. All interested Veterans will be consented and enrolled into the study prior to the pre-screening interview and Veterans that fit into the selected groups for the MRI study will receive a separate invitation to participate in that arm of the study. The five groups of Veterans that will be required to complete this study are described below.

* Current WBV Group (Group 1) will consist of Veterans with no history of active duty occupational WBV exposure, but with civilian occupational WBV exposure as a Veteran. These individuals will be less than 45 years old and have less than 5 years of civilian occupational WBV exposure. This group will demonstrate the effects of civilian occupational WBV exposure on endplate degeneration, IVD fluid dynamics, and spine structural degeneration metrics. Three multi-parametric MRI scans obtained over the course of this four-year protocol (aim 1) will allow for tracking of endplate health and identification of progressive changes in spine structural characteristics such as lumbar Cobb angle, disc/foraminal dimensions, endplate degeneration, and intervertebral disc perfusion and hydration. These changes will be correlated with WBV logs maintained by each enrolled subject that will provide weekly estimates of the type and duration of occupational exposure over the duration of the study. An experimental acute WBV protocol (aim 2) will outline the acute response of the lumbar spine endplates and intervertebral discs to WBV This protocol will consist of a baseline upright MRI scan in the morning, 30 minutes of experimental WBV, and a second post-WBV upright MRI scan in the afternoon. Subjects will be selected for participation in the MRI arm of the study to ensure consistency in occupational WBV characteristics (e.g., heavy equipment operators versus long haul truck drivers) and duration of occupation to reduce the variability in ongoing occupational WBV that may influence the current spine health at the time of enrollment
* Military WBV Group (Group 2) will consist of Veterans with at least 6 years of active duty WBV exposure (ex. heavy equipment operators, helicopter pilots, small watercraft operators). These individuals will be less than 45 years old and have no civilian occupational exposure to WBV. This group will undergo two series of supine multi-parametric MRI scans at the beginning and end of the study (aim 1) and the experimental acute WBV protocol as described above (aim 2). Our pre-screening process will allow us to select a group of individuals that had similar active duty WBV characteristics in terms of type and duration of occupation. Subjects will be selected for participation in the MRI arm of the study to ensure consistency in Military WBV characteristics (e.g., helicopter pilots versus fast boat drivers) and duration of military occupation to reduce the variability in WBV history that may influence the current spine health at the time of enrollment.
* No WBV Group (Control Group) (Group 3) will consist of Veterans with no history of active duty or civilian occupational exposure to WBV. These individuals will be age and sex matched with Current WBV and Military WBV Groups and will not experience any fluid restriction. This group will undergo the same procedures as the Current WBV Group, including three multi-parametric MRI scans (aim 1) and one exposure to the acute WBV protocol (aim 2).
* Hydrated Group (Group 4). The No WBV Group from aims 1 and 2 of the study will participate in aim 3, participating in multi-parametric MRI scans in both a well hydrated state and a dehydrated state. A 3-day fluid log will be maintained following consent to provide a fluid intake baseline. The 3 days prior to their arrival participants will be asked to consume at least 2.7 liters (11 cups) of fluids per day for female participants, and at least 3.7 liters (16 cups) for male participants. Hydration status will be confirmed with measurements of urine specific gravity values less than 1.010. The day prior to multi-parametric MRI scanning, participants will be asked to refrain from rigorous exercise. This group will participate in the Hydrated MRI protocol during Year 3 of the study.
* Dehydrated Group (Group 5). The No WBV Group from aims 1 and 2 of the study will participate in aim 3, participating in multi-parametric MRI scans in both a well hydrated state and a dehydrated state. A 3-day fluid log will be maintained following consent to provide a fluid intake baseline. The 3 days prior to their arrival participants will be asked to consume about 1.3 liters (5.5 cups) of fluids per day for female participants, and about 1.8 liters (8 cups) for male participants. Hydration status will be confirmed with measurements of urine specific gravity values greater than 1.020. The day prior to multi-parametric MRI scanning, participants will be asked to refrain from rigorous exercise. This group will participate in the Dehydrated MRI protocol during Year 4 of the study.

Veterans selected for the MRI arm of the study will be informed of this decision via a letter that will describe their study group, the MRI procedures in which they will be asked to participate, their study-specific subject number, and their stipend for participation. They must then agree to participate by signing and returning an included consent form to the study team. After they have agreed to participate in the MRI arm of the study, a study team member will work with them to schedule their MRI scan(s) at either MCW Center for Imaging Research (supine scans) or Upright MRI of Deerfield (Upright scans), depending on their study group. Veterans will then be provided with information on the date/time of their scan, when to arrive, facility and parking locations (including map), how long the scan will take, what they should wear, and any fluid restrictions if necessary. They will be informed that a study team member will meet them at the scan location, prior to their scan, and will guide them through the process. Veterans will also be informed that they have been given a study-specific de-identified subject number to ensure their privacy and that they can use that number to identify themselves the study team member and the MRI facility upon arrival.

Veterans will be responsible for their own transport to the MRI facility. Upon arrival, they will be met at the facility by a study team member. The study team member will confirm their study-specific subject number, describe the procedures that will occur, how long the entire process will take, and answer any questions that the Veteran may have. Veterans will be asked to arrive at the MRI facility approximately 30 minutes prior to their MRI scan time. If the Veteran is not wearing MRI appropriate clothing, they will be guided to a changing room where they can change into scrubs provided by the facility. Prior to scanning, Veterans will be asked to fill out an MRI screening form that will ask MRI-relevant questions regarding implants and medical conditions. The MRI screening form is included as a part of this IRB submission.

Each MRI scan will last no more than 60 minutes. Participation in Aim 1 will include a total of three MRI scans; the first MRI scan in Year 1 of the study, the second in Years 2 or 3, and the third in year 4. Participation in Aims 2 and 3 will include 2 MRI scans and one whole body vibration protocol on the same day. The whole body vibration protocol will consist of the following. Acute whole body vibration will be delivered through a low backed chair mounted on a controlled vibrating platform. Participants will experience a 30-minute vertical vibration session of 5 Hz with a peak-to-peak amplitude of 3 mm, and a peak acceleration of 2 m/s2. This exposure was used previously, determined to be safe for participants, and was shown to have a measurable effect on diurnal height changes [Sullivan Spine 1990].

Urine samples will be collected prior to MRI scans for Hydrated and Dehydrated groups in Aim 3. Upon arrival at the MRI facility, each subject will be provided with a urine collection container by the Study Team member, who will describe the "clean-catch" method for collection. That method involves starting to urinate, stopping, collecting urine mid-stream in the container, then finishing urination in the toilet. The subject will then give the contained back to the Study Team member, who will place it in a refrigerated container. Following the MRI scan, the Study Team member will return the same to our labs at the ZVAMC and analyze specific gravity of the sample using a refractometer.

Recruitment Aim 1 has a total of 3 experimental groups (Current WBV, Military WBV, and No WBV), and three MRIs per subject. 39 subjects (13 per group) are required, who will undergo a total of 117 supine MRIs.

Aim 2 has a total of 3 experimental groups (Current WBV, Military WBV, and No WBV), and two upright MRIs per subject. 39 subjects (13 per group) are required, for a total of 78 upright MRIs. However we feel that the effect size for this experiment will be higher than the effect size in the preliminary data since the proposed experiment will measure acute mechanically-induced changes in disc hydration following WBV, whereas groupwise differences in our preliminary data were the result of chronic degenerative changes in disc hydration.

Therefore, we anticipate having the ability to detect statistically significant and appropriately powered groupwise differences during this experiment, even with smaller group sizes.

Aim 3 has a total of 2 experimental groups (hydrated and dehydrated), and two MRIs per subject. 34 subjects (17 per group) are required, who will undergo a total of 68 MRIs.

Potential research subjects will be identified using VA Informatics and Computing Infrastructure (VINCI). All potential subjects will be notified via letter that they meet the preliminary requirements for inclusion in a research study being conducted by Investigators at the ZVAMC. They will be asked to respond via telephone or email if interested and notified that we will follow up with a phone call approximately two weeks after the date of the letter to confirm whether they would like to participate. This protocol is common for other human studies at ZVAMC and has been in use by our Translational Research Unit (TRU) for years. All interested Veterans will be interviewed at a time of their choosing via telephone or in person interviews to determine their suitability for inclusion in this study.

Veterans that consent for initial enrollment will be provided with baseline questionnaires about military service, current and prior whole body vibration exposure, pain intensity, pain-related disability, and modifiers of pain, using the questionnaires listed below. Study team members will review the list of Veterans that have agreed to the initial enrollment on an ongoing basis. We will stop enrolling new subjects when we have obtained a sufficient number for matched cohorts for each experimental group based on similarity in age, whole body vibration characteristics, and pain profile.

Subjects from each matched cohort will be asked to participate in Aims 1 and 2 (Groups 1, 2, and 3) or Aim 3 (additional Group 3 enrollment). Aims 1 and 2 will enroll 39 subjects (13 per group for Groups 1, 2, and 3) that will receive a total of 5 MRI scans (3 at MCW and 2 at Upright MRI of Deerfield). Aim 3 will enroll an additional 34 subjects (17 per group x 2 groups) that will each receive 2 MRI scans at MCW. This will result in a minimum of 73 ZVAMC Veterans (13 per group x 3 groups for Aims 1 and 2; 17 per group x 2 groups for Aim 3) enrolled in the study. However, we anticipate that some subjects may not be willing to participate in multiple arms of the study. Since each Aim includes repeated measurements so that subjects can be used as their own controls, the study protocol will allow for separate cohorts of Veterans to be enrolled in each Aim. Therefore, the maximum enrollment for the study, if we had separate cohorts for each Aim, would be 112 Veterans (39 for Aim 1, 39 for Aim 2, 34 for Aim 3).

ELIGIBILITY:
Inclusion Criteria:

* English speaking; Male/Female Veterans age 20-45 years; BMI < 30; ability to sit upright for 60 mins; ability to drive to Deerfield, IL; ambulatory

Exclusion Criteria:

* Previous spinal surgery; conditions/diseases associated with altered pain perception including neurological diseases (e.g., multiple sclerosis, trigeminal neuralgia, central sensitization), major psychiatric disorders, diabetes, neoplasm and cardiovascular disorders, chronic widespread pain diagnosis, pregnant women, MRI contraindications.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Occupational Whole Body Vibration History | Whole body vibration questionnaires will be provided at the time of enrollment and immediately prior to each MRI scan.
  We will use questionnaires to quantify each subject's history with regard to occupational whole body vibration. Groups will include subjects that had whole body vibration while in the military, subjects that have current occupations with whole body vibration, and subjects that have not significant history of whole body vibration.
Oswestry Disability Index | ODI will be collected at the time of enrollment and again immediately prior to each MRI scan.
  Patient-reported outcome measure that assesses the degree to which low back pain impacts a person's daily functioning. The questionnaire consists of 10 sections (pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life, traveling). Each section has 6 statements scored 0-5; patient selects the statement that best describes them.

CONTACTS AND LOCATIONS:
Overall Officials: Brian D Stemper, PhD, Principal Investigator — Milwaukee VA Medical Center
Locations (1):
- Zablocki Veterans Affairs Medical Center, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Written requests for IPD must be made directly to the study PI. The request must include a description of the specific data being requested, the purpose for the request, anticipated outcomes from usage of IPD, and a statement that the study and PI will be acknowledged in any publications resulting from use of IPD. The Investigative Team will evaluate any requests and will decide to share or not share IPD. Only de-identified data will be provided.
Supporting Information: Study Protocol, ICF
Time Frame: The Study Team will review requests for IPD following the first year of the study and will continue reviewing requests indefinitely.
Access Criteria: The Study Team will evaluate each request individually and decide on the type and format of data that will be shared.